CLINICAL TRIAL: NCT02372253
Title: Repurposing of Verapamil as a Beta Cell Survival Therapy in Type 1 Diabetes
Brief Title: Verapamil for Beta Cell Survival Therapy in Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Fernando Ovalle, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3-SRA-2014-302-M-R
Record Dates: First submitted 2015-02-20; First posted 2015-02-26 (Estimated); Results first posted 2019-01-30 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2019-01

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: verapamil; type 1 diabetes; diabetes; beta cells; beta cell function; insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance | interventions — Verapamil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Verapamil (Experimental): 13-26 subjects with Type 1 Diabetes meeting the inclusion criteria will be randomly assigned to receive daily oral verapamil for 12 months. The initial dose of verapamil will be 120 mg daily, and this will be advanced if tolerated to a maximum dose of 360 mg daily. The verapamil tablets will be encapsulated to match the placebo capsules
  Interventions: Drug: Verapamil
- Placebo (Placebo Comparator): 13-26 subjects with Type 1 Diabetes meeting the inclusion criteria will be randomly assigned to receive daily oral placebo for 12 months. The initial dose of placebo will be 120 mg daily, and this will be advanced if tolerated to a maximum dose of 360 mg daily. The placebo tablets will be encapsulated to match the verapamil capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Verapamil
  Arms: Verapamil
Drug: Placebo
  Arms: Placebo

SUMMARY:
The overall purpose of this trial is to assess the efficacy and safety of using oral verapamil in subjects with recent onset T1D in order to downregulate TXNIP and enhance the patients' endogenous beta cell mass and insulin production. The objectives are therefore to assess parameters of beta cell survival (including new biomarkers), insulin production and glucose control and the feasibility of this approach and thereby provide the basis for future, larger/expanded, longer-term verapamil studies and the off-label use of this approved drug for Type 1 Diabetes (T1D).

DETAILED DESCRIPTION:
Loss of pancreatic beta-cell mass is a key factor in T1D, but therapies to halt this process are not available. The investigators have discovered thioredoxin-interacting protein (TXNIP), as a promising target in this regard and have now found that the commonly used anti-hypertensive drug and calcium channel-blocker, verapamil, effectively lowers beta-cell TXNIP expression in rodent beta-cells and human islets, promotes beta-cell survival and rescues mice from T1D. This makes verapamil a potentially attractive drug for T1D, but prospective clinical data are lacking. The investigators primary objective is therefore to conduct a randomized, placebo-controlled, double-blind study of the efficacy and safety of verapamil in adults with recent-onset T1D and to demonstrate that subjects on oral verapamil daily for 12 months will have improved insulin production (as an indirect measure of beta-cell mass).

Results will have major translational implications with potential immediate impact on clinical care, encourage large clinical follow-up trials, evaluate markers of beta cell health and ultimately help develop a novel therapy that enhances the patient's own beta-cell mass and function.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following criteria:
* Diagnosis of Type 1a Diabetes Mellitus based on American Diabetes Association (ADA) Criteria
* Written informed consent obtained from the subject including consent for the use of research-related health information
* ≥ 18 years of age and ≤ 45 years of age
* < 3 months since T1D was diagnosed
* BMI < 30
* Baseline A1c <10%
* Detectable fasting or stimulated C-peptide level (above the lower limit of detection of the assay)
* C-peptide increase during screening mixed meal tolerance test with a minimal stimulated value of ≥ 0.2 pmol/mL
* Presence of antibodies to at least one of the following antigens: insulin, glutamic acid decarboxylase (GAD)-65, Insulinoma Antigen 2 (IA-2) and Zinc Transporter 8 (ZnT8)
* Agree to intensive management of diabetes with a HgbA1c goal of < 7.0% and willing to wear and insulin pump and Continuous Glucose Monitoring System (CGMS)
* If female, (a) surgically sterile or (b) postmenopausal or (c) if of reproductive potential, willing to use medically acceptable birth control (e.g. female hormonal contraception, barrier methods or sterilization) until 3 months after completion of any Treatment Period
* Serum creatinine ≤ 1.5 x upper limit of normal (ULN)
* Currently receiving insulin therapy
* Willing to forego other forms of experimental treatment during the study

Exclusion Criteria:

* Subjects must have none of the following:
* Any medical condition that, in the opinion of the investigator, would interfere with safe completion of the trial
* Pregnant females or lactating females who intend to provide their own breast milk to the baby during the study
* Current therapy with Glucagon-like peptide (GLP)-1 receptor agonists, pramlintide, or any other agents that might be thought to potentially stimulate pancreatic beta cell regeneration or insulin secretion
* Current treatment with oral antidiabetic agents
* Uncompensated heart failure, fluid overload, myocardial infarction or evidence of ischemic heart disease or other serious cardiac disease as described in New York Heart Association (NYHA) Class III or IV criteria within the 12 weeks before randomization
* History of epilepsy, cancer, cystic fibrosis, sickle cell anemia, neuropathy, peripheral vascular disease or cerebrovascular disease
* Untreated hypothyroidism or active Graves' disease with hyperthyroidism
* Treatment with systemic glucocorticoid therapy by oral, intravenous (IV), or intramuscular (IM) route within 12 weeks before randomization; patients who are likely to require treatment with corticosteroids during the trial are also excluded
* Evidence of active infection
* Total bilirubin > 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 1.5 x ULN
* A psychiatric or medical disorder that would prevent giving informed consent
* Hypersensitivity to verapamil or any component of the formulation; known left ventricular dysfunction; hypotension (systolic pressure <90 mm Hg); PR interval prolongation on EKG or any bradyarrhythmia (e.g. sick sinus syndrome, Anterior Ventral (AV) block); atrial flutter or fibrillation, and an accessory bypass tract (Wolff-Parkinson- White (WPW) syndrome, Lown-Ganong-Levine syndrome)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-02; Primary Completion 2017-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Ovalle, MD, Principal Investigator — University of Alabama at Birmingham; Anath Shalev, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 32 subjects with recent-onset Type 1 diabetes were screened for autoantibodies and MMTT-stimulated C-peptide. Five were not eligible for randomization (3 were antibody negative and 2 were C-peptide negative). One additional participant declined.
Groups:
- Verapamil: Verapamil Sustained Release (SR) 360mg Daily
- Placebo: Matching Placebo
Period: Overall Study
Arm/Group | Verapamil | Placebo
Started | 13 | 13
Completed | 11 | 13
Not Completed | 2 | 0
Not completed — Non Compliance | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Verapamil: Verapamil SR 360mg Daily
- Total: Total of all reporting groups
Arm/Group | Verapamil | Placebo | Total
Number analyzed (Participants) | 11 | 13 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (2.3) | 28.3 (2.1) | 30.3 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 6 | 8 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 10 | 13 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 13 | 24
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.4 (0.8) | 22.1 (0.7) | 23.25 (0.75)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mmol/L] | 6.4 (1) | 6.9 (1) | 6.65 (1)
HbA1C [Mean (Standard Deviation); unit: %] | 6.6 (0.4) | 6.8 (0.3) | 6.7 (0.4)

OUTCOME MEASURES:

1. Primary Outcome: Functional Beta Cell Mass
Description: Functional Beta Cell Mass as determined by the area under the curve (AUC) from a 2-hour Mixed Meal-Stimulated C-peptide after daily verapamil for 12 months. A greater improvement in insulin production (as an indirect measure of beta cell mass) in subjects receiving verapamil as compared to those receiving placebo would provide an indication of the efficacy of this intervention. The C-peptide AUC (0-120 min) was calculated by using the trapezoidal rule and was divided by the time of the test to obtain the mean AUC (in nmol/L).
Time Frame: 12 months
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Verapamil | Placebo
Number analyzed (Participants) | 11 | 13
nmol/L | 0.74 (0.07) | 0.46 (0.08)

2. Secondary Outcome: Percent Change From Baseline in Exogenous Insulin Requirements
Description: Percent change in exogenous insulin requirements over the last 7-14 consecutive days at 12 months. This will be assessed as a surrogate inverse marker of residual beta cell function.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | Verapamil | Placebo
Number analyzed (Participants) | 11 | 13
Percent Change | 27.0 (15.6) | 69.8 (7.9)

3. Secondary Outcome: Percent Change From Baseline in Exogenous Insulin Requirements
Description: Percent change in exogenous insulin requirements over the last 7-14 consecutive days at 12 weeks. This will be assessed as a surrogate inverse marker of residual beta cell function.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | Verapamil | Placebo
Number analyzed (Participants) | 11 | 13
Percent Change | 5.9 (11.4) | 26.0 (9.5)

4. Secondary Outcome: HbA1C
Description: Glycemic control, as measured by HbA1c. In addition to being an important determinant of residual beta cell function/survival, it also helps reveal a more complete picture of beta cell function.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Verapamil | Placebo
Number analyzed (Participants) | 11 | 13
Percent | 6.4 (0.2) | 6.9 (0.3)

5. Secondary Outcome: HbA1c
Description: as for outcome 4
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Verapamil | Placebo
Number analyzed (Participants) | 11 | 13
Percent | 6.0 (0.1) | 6.6 (0.3)

6. Secondary Outcome: Hypoglycemic Events
Description: Glycemic control, as measured by hypoglycemic events.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: events per month
Groups:
- Verapamil: 13-26 subjects with Type 1 Diabetes meeting the inclusion criteria will be randomly assigned to receive daily oral verapamil for 12 months. The initial dose of verapamil will be 120 mg daily, and this will be advanced if tolerated to a maximum dose of 360 mg daily. The verapamil tablets will be encapsulated to match the placebo capsules
  Verapamil
- Placebo: 13-26 subjects with Type 1 Diabetes meeting the inclusion criteria will be randomly assigned to receive daily oral placebo for 12 months. The initial dose of placebo will be 120 mg daily, and this will be advanced if tolerated to a maximum dose of 360 mg daily. The placebo tablets will be encapsulated to match the verapamil capsules
  Placebo
Arm/Group | Verapamil | Placebo
Number analyzed (Participants) | 11 | 13
events per month | 0.55 (0.31) | 2.72 (0.86)

7. Other Pre Specified Outcome: Beta Cell Markers
Description: Beta cell markers. We will collect serum at baseline and at Week 12 and Months 6, 9 and 12 for future assessment of putative beta cell markers.
Time Frame: 12 weeks and 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the 1 year subjects received study treatment.
Arm/Group | Verapamil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/13
Other Adverse Events (participants affected / at risk) | 7/11 | 2/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Verapamil (N=11) | Placebo (N=13)
Constipation (Gastrointestinal disorders) | 5 (5) | 1 (1)
Dizziness (General disorders) | 1 (1) | 0 (0)
Nausea (General disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT02372253/Prot_SAP_000.pdf